CLINICAL TRIAL: NCT05870813
Title: Cancer Landscape - Early Adjuvant Retrospective Registry - Breast Cancer (CLEAR-B)
Brief Title: CLEAR-B: Cancer Landscape - Early Adjuvant Retrospective Registry - Breast Cancer
Acronym: CLEAR-B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut fuer Frauengesundheit (Other)
Collaborators: AGO Breast Study Group e.V. (Unknown); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: IFG-02-2022; AGOB-059 (Other: AGO breast study group)
Record Dates: First submitted 2023-04-14; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; HER2-negative Breast Cancer; Hormone Receptor Positive Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AI+OFS: adjuvant treatment with aromatase inhibitor + OFS (ovarian function suppression)
- TAM: Patients started the adjuvant treatment with Tamoxifen ± OFS

SUMMARY:
This is a non-interventional retrospective cohort study of premenopausal patients with HR+/HER2- breast cancer who are treated in the adjuvant setting with either Tamoxifen, Tamoxifen + Ovarial Function Suppression or Aromatase inhibitor + Ovarial Function Suppression.

DETAILED DESCRIPTION:
The treatment landscape concerning the adjuvant endocrine therapy in premenopausal patients with early-stage hormone receptor positive (HRpos) breast cancer is quite heterogeneous and therapy recommendations can vary. Tamoxifen (TAM) is a common treatment option that does not require OFS, but research suggests that adding OFS to tamoxifen may improve outcomes. Aromatase inhibitors (AI) are another option, but they can only be used with OFS for premenopausal patients. Studies have shown that AI + OFS improves disease-free survival compared to TAM + OFS, but it may lead to additional side effects such as osteopenia and bone fractures.

The CLEAR-B study aims to provide a detailed description of the therapy landscape in this therapeutic setting, including recurrence rates and overall survival with AI compared to TAM, as well as a comparison of the chosen therapies within prognostic subgroups.

CLEAR-B is a retrospective cohort study, collecting data of premenopausal patients who were diagnosed with early-stage breast cancer between January 2016 and June 2019 in a certified breast cancer center. These patients had an intermediate or high risk of cancer recurrence, as defined by (neo)adjuvant chemotherapy, and/or pT≥2cm at the timepoint of definitive surgery and/or at least one positive lymph node at the time of definite surgery (pN+).

The primary objective is to compare the invasive disease-free survival (iDFS) of patients who were treated with AI + OFS vs. those who were treated with TAM ± OFS. Additionally, the study will compare distant disease-free survival (DDFS) and overall survival (OS) between the two groups and perform subgroup analyses according to risk stratification (stage II and III). This study will be conducted at around 75 certified breast cancer centers and will enroll up to 3000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with a first primary diagnosis of hormone receptor-positive, HER2- negative unilateral early breast cancer for whom an endocrine treatment is indicated
* Patients must be at least 18 years of age but not older than 60
* Premenopausal defined as all statements must be true

  * No oophorectomy before the diagnosis of breast cancer
  * Women with uterus: Regular, physiological menses at the timepoint of therapy decision for anti-endocrine treatment in the absence of contraceptives and hormonal treatment
  * Women without uterus and remaining ovaries: premenopausal hormone levels must be documented at the time of therapy decision for anti-endocrine treatment
* Patients with an intermediate or high-risk early-stage breast cancer defined as: At least one of the following must be fulfilled

  * (Neo)adjuvant chemotherapy
  * pT≥2cm at the timepoint of definitive surgery
  * at least one positive lymph node at the time of definite surgery (pN+)
* Patient must be previously registered in and must have been documented as part of the certification process for a certified breast cancer center according to the Deutsche Krebsgesellschaft/Deutsche Gesellschaft für Senologie
* Breast Cancer must have been diagnosed between Jan 2016 and Jun 2019

Exclusion Criteria:

* Patients with a low recurrence risk (see inclusion criteria for definition)
* Locally advanced breast cancer or distant metastases at diagnosis
* Male biological sex
* Patients not treated in a certified breast cancer center
* Treatment with CDK4/6Previous diagnosis of invasive breast cancer or in situ breast cancer
* Concurrent invasive malignancy
* Bilateral breast cancer at the timepoint of diagnosis
* Previous diagnosis of invasive breast cancer or in situ breast cancer is not allowed

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Premenopausal patients with early-stage breast cancer who have been diagnosed from January 2016 to June 2019 with an intermediate or high recurrence risk in a certified breast cancer center (DKG/DGS).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
iDFS | First start of adjuvant endocrine therapy until date of the above mentioned events up to 5 years
  The primary study aim is to show that aromatase inhibitor (AI) based treatments (AI arm) are not inferior to treatments based on tamoxifen (tamoxifen arm) in terms of invasive diseasefree survival (iDFS).
  iDFS will be assessed as time to event. Events for iDFS include: Invasive Ipsilateral Breast Tumor Recurrence (IBTR), Local/Regional Invasive Recurrence, Distant Recurrence, Death from BC, Death from Non-BC Cause, Death From unknown cause, Invasive Contralateral BC, Second Primary Invasive Cancer (non-breast)
Comparison of iDFS | First start of adjuvant endocrine therapy until date of the above mentioned events up to 5 years
  In case non-inferiority is confirmed, the superiority of Cohort AI+OFS over Cohort TAM will be tested with regard to iDFS.
  iDFS will be assessed as time to event. Events for iDFS include: Invasive Ipsilateral Breast Tumor Recurrence (IBTR), Local/Regional Invasive Recurrence, Distant Recurrence, Death from BC, Death from Non-BC Cause, Death From unknown cause, Invasive Contralateral BC, Second Primary Invasive Cancer (non-breast)

SECONDARY OUTCOMES:
Comparison of DDFS | First start of adjuvant endocrine therapy until date of the above mentioned events up to 5 years
  To analyze the non-inferiority of the Cohort AI+OFS compared with the Cohort TAM with regard to distant disease-free survival (DDFS). DDFS will be assessed as time to event. Events for DDFS include distant recurrence, death from breast cancer, death from non-breast cancer cause, death from unknown cause.
Comparison of OS | First start of adjuvant endocrine therapy until date of death up to 5 years
  To analyze the non-inferiority of the Cohort AI+OFS compared with the Cohort TAM with regard to overall survival (OS). In case non-inferiority is confirmed, the superiority of Cohort AI+OFS over Cohort TAM will be tested with regard to OS.
  OS is defined as time from first start of adjuvant endocrine therapy until date of death due to any cause.
Comparison of iDFS in Cohort TAM | First start of adjuvant endocrine therapy until date of the above mentioned events up to 5 years
  To compare patients within the Cohort TAM who were treated with OFS and those who were not treated with OFS. iDFS will be assessed as time to event. Events for iDFS include: Invasive Ipsilateral Breast Tumor Recurrence (IBTR), Local/Regional Invasive Recurrence, Distant Recurrence, Death from BC, Death from Non-BC Cause, Death From unknown cause, Invasive Contralateral BC, Second Primary Invasive Cancer (non-breast)
Comparison of DDFS in Cohort TAM | First start of adjuvant endocrine therapy until date of the above mentioned events up to 5 years
  To compare patients within the Cohort TAM who were treated with OFS and those who were not treated with OFS. DDFS will be assessed as time to event. Events for DDFS include distant recurrence, death from breast cancer, death from non-breast cancer cause, death from unknown cause.
Comparison of OS in Cohort TAM | First start of adjuvant endocrine therapy until date of death up to 5 years
  To compare patients within the Cohort TAM who were treated with OFS and those who were not treated with OFS. OS is defined as time from first start of adjuvant endocrine therapy until date of death due to any cause.
Comparison of iDFS (TAM+OFS and AI+OFS) | First start of adjuvant endocrine therapy until date of the above mentioned events up to 5 years
  To compare patients of Cohort AI+OFS with patients in Cohort TAM, who were treated with OFS with regard to iDFS.
  iDFS will be assessed as time to event. Events for iDFS include: Invasive Ipsilateral Breast Tumor Recurrence (IBTR), Local/Regional Invasive Recurrence, Distant Recurrence, Death from BC, Death from Non-BC Cause, Death From unknown cause, Invasive Contralateral BC, Second Primary Invasive Cancer (non-breast)
Comparison of DDFS (TAM+OFS and AI+OFS) | First start of adjuvant endocrine therapy until date of the above mentioned events up to 5 years
  To compare patients of Cohort AI+OFS with patients in Cohort TAM, who were treated with OFS with regard to DDFS. DDFS will be assessed as time to event. Events for DDFS include distant recurrence, death from breast cancer, death from non-breast cancer cause, death from unknown cause.
Comparison of OS (TAM+OFS and AI+OFS) | First start of adjuvant endocrine therapy until date of death up to 5 years
  To compare patients of Cohort AI+OFS with patients in Cohort TAM who were treated with OFS.
  OS is defined as time from first start of adjuvant endocrine therapy until date of death due to any cause.
Comparison of iDFS (TAM-OFS and AI+OFS) | First start of adjuvant endocrine therapy until date of the above mentioned events up to 5 years
  To compare patients of Cohort AI+OFS with patients in Cohort TAM, who were not treated with OFS with regard to iDFS.
  iDFS will be assessed as time to event. Events for iDFS include: Invasive Ipsilateral Breast Tumor Recurrence (IBTR), Local/Regional Invasive Recurrence, Distant Recurrence, Death from BC, Death from Non-BC Cause, Death From unknown cause, Invasive Contralateral BC, Second Primary Invasive Cancer (non-breast)
Comparison of DDFS (TAM-OFS and AI+OFS) | First start of adjuvant endocrine therapy until date of the above mentioned events up to 5 years
  To compare patients of Cohort AI+OFS with patients in Cohort TAM, who were not treated with OFS with regard to DDFS.
  DDFS will be assessed as time to event. Events for DDFS include distant recurrence, death from breast cancer, death from non-breast cancer cause, death from unknown cause.
Comparison of OS (TAM-OFS and AI+OFS) | First start of adjuvant endocrine therapy until date of death up to 5 years
  To compare patients of Cohort AI+OFS with patients in Cohort TAM who were not treated with OFS.
  OS is defined as time from first start of adjuvant endocrine therapy until date of death due to any cause.
Influence of disease stage | Baseline until onset of disease progression or death up to 5 years
  To conduct multivariate analyses to estimate the influence of disease stage on prognosis.
Risk Factors | Baseline until onset of disease progression or death up to 5 years
  To conduct subgroup analyses for the survival outcomes (iDFS, DDFS, OS) according to risk stratification (stage II and stage III)
NATALEE Comparison | Baseline until onset of disease progression or death up to 5 years
  To compare patients who are matching the inclusion and exclusion criteria of the pivotal study NATALEE and who were treated in Cohort AI+OFS with patients matching the NATALEE population and who were treated in Cohort TAM.

OTHER OUTCOMES:
Therapy frequencies | Baseline
  To assess the frequency of the different therapies according to risk groups
Adherence | End of Treatment/ Treatment termination up to 5 years
  Number of patients with specified reason for therapy termination (recurrence, side effects, patients' wishes etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecology and Obstetrics, Erlangen University Hospital, Erlangen, Germany